CLINICAL TRIAL: NCT06093945
Title: Study to Evaluate the Drug-drug Interaction Effect of Omeprazole on the Pharmacokinetics of SHR2554 in Healthy Subjects: A Single-center, Open-label, Single-dose, Two-period, Fixed Sequence, Self-controlled Study
Brief Title: Effect of Omeprazole on Pharmacokinetics of SHR2554 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-112
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose, two-period, fixed sequence, self-controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR2554 and omeprazole (Experimental): Sequential treatments of SHR2554 alone followed by SHR2554+ omeprazole, with a washout period in between.
  Interventions: Drug: SHR2554 tablet dosing; Drug: Omeprazole tablet dosing

INTERVENTIONS:
Drug: SHR2554 tablet dosing — SHR2554 350mg taken on Day 1 and Day 10
Drug: Omeprazole tablet dosing — Omeprazole taken from Days 5 to Day 10

SUMMARY:
The study aimed to assess the effects of omeprazole on single-dose SHR2554 in healthy subjects, exploring the pharmacokinetic changes of SHR2554 and ensuring the safety when SHR2554 is co-administered with omeprazole.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form before the trial and have a full understanding of the trial's content, procedures, and potential adverse reactions.
2. Be able to complete the study according to the trial protocol.
3. Healthy male and female subjects aged 18 to 45 (inclusive) on the day of signing the informed consent form.
4. Female subjects of childbearing potential must use effective contraception for 1 month from the date of signing the informed consent form until the last dose. Serum HCG testing before dosing must be negative. Male subjects with partners of childbearing potential must agree to use effective contraception measures and avoid sperm donation during the trial and for 1 month after the last administration of SHR2554.
5. Male subjects must weigh at least 50 kg, and female subjects must weigh at least 45 kg, with a body mass index (BMI) ranging from 19 kg/m2 to 26 kg/m2 (inclusive).
6. Health Condition: No history of heart, liver, kidney, gastrointestinal, neurological, psychiatric abnormalities, or metabolic disorders.
7. Normal or clinically insignificant findings in vital signs, physical examination, routine laboratory tests (complete blood count, blood biochemistry, urinalysis, coagulation function, myocardial enzyme profile, thyroid function), echocardiography, posteroanterior chest X-ray, and abdominal ultrasound.
8. Fridericia-corrected QT interval (QTcF) of males should ≤ 430 ms, and ≤ 450 ms for females. Left ventricular ejection fraction (LVEF) should ≥ 50%.

Exclusion Criteria:

1. Positive results on screening tests for hepatitis B surface antigen, hepatitis C antibodies, syphilis spirochete antibodies, or HIV antibodies.
2. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to SHR2554, its excipients, or drugs with a similar chemical structure or class.
3. Poorly controlled clinical heart symptoms or diseases such as: (1) NYHA Class 2 or higher heart failure; (2) Unstable angina; (3) Myocardial infarction within the past year; (4) Any supraventricular or ventricular arrhythmia requiring treatment or intervention.
4. Occurrence of any of the following conditions within the past 6 months before screening: Myocardial infarction, severe/unstable angina, NYHA Class II-IV heart failure, continuous arrhythmias of ≥ Grade 2 (graded based on NCI CTCAE 5.0), heart failure, second or third-degree atrioventricular block, complete left bundle branch block, any grade of atrial fibrillation, coronary/peripheral artery bypass grafting or stent implantation, cerebrovascular accident (including transient ischemic attack), pulmonary embolism, deep vein thrombosis.
5. Use of any medication within the 4 weeks prior to the initial dose that carries a risk of prolonged QT/QTc interval or causing torsades de pointes (TdP) arrhythmia; a history of congenital QT interval prolongation syndrome or a family history of QT interval prolongation; presence of an implanted pacemaker or automated implantable cardioverter-defibrillator; uncorrected electrolyte disturbances, or any factors affecting QT/QTc studies.
6. Pulmonary diseases, including infiltrative lung diseases, pneumonia, and respiratory distress.
7. Chronic kidney disease, renal insufficiency, or a history of renal anemia.
8. History of difficulty swallowing or any gastrointestinal disorders that affect drug absorption.
9. Any uncontrolled digestive ulcers, colitis, pancreatitis, etc.
10. Other primary diseases of important organs, such as neurological, cardiovascular, urological, digestive, respiratory, metabolic, and musculoskeletal system disorders, which makes the investigator believes it is unsuitable for participation in this study.
11. Subjects who have undergone any surgery within 3 months prior to screening that could affect drug absorption, distribution, metabolism, or elimination.
12. Subjects who have undergone any surgery within 6 months prior to screening.
13. Subjects who have taken hepatotoxic drugs (such as acetaminophen, erythromycin, fluconazole, ketoconazole, rifampin, etc.) within 6 months prior to screening.
14. Subjects who have participated in a clinical trial within 3 months prior to screening.
15. Subjects who have taken known CYP3A or CYP2C19 inducers/inhibitors (see Appendices 2 and 3) within 28 days prior to the first administration of SHR2554.
16. Subjects who have taken any prescription or non-prescription medications within 7 days prior to the first administration of SHR2554.
17. Subjects who have consumed any vitamin products or herbal supplements within 7 days prior to the first administration of SHR2554.
18. Subjects who abuse alcohol or excessive intake of alcohol within 6 months prior to screening, defined as consuming more than 14 units of alcohol per week (1 unit = 285 mL of beer, 25 mL of 40% alcohol, or 100 mL of wine); or subjects with an alcohol breath test result ≥20 mg/dL during screening.
19. Subjects who have smoked more than 5 cigarettes per day or habitually use nicotine-containing products within 3 months prior to screening, and are unable to quit during the study or have a positive nicotine screening result during screening.
20. Subjects who misuse drugs or have used recreational drugs (such as cannabis) within 3 months prior to screening, or have used hard drugs (such as cocaine, amphetamines, ecstasy, etc.) within the past year, or have a positive result on drug abuse (substance abuse) screening during screening.
21. Subjects who have consumed grapefruit or grapefruit-containing products, caffeine, xanthine, or alcohol-containing foods or beverages within 48 hours prior to the first administration of SHR2554; engaged in strenuous exercise, or have other factors that may affect drug absorption, distribution, metabolism, or excretion.
22. Subjects who habitually consume grapefruit juice or excessive amounts of tea, coffee, and/or caffeinated beverages, and are unable to abstain during the study.
23. Subjects who donated blood within the last 3 months and donated ≥400 mL of blood or experienced blood loss ≥400 mL, donated blood within the last 1 month and donated ≥200 mL of blood or experienced blood loss ≥200 mL, or received a blood transfusion.
24. Subjects with a history of syncope or vasovagal episodes, difficulty with blood collection, or an inability to tolerate venipuncture.
25. Subjects who, in the opinion of the investigator, have other factors that make them unsuitable for participation in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Cmax of SHR2554: Rate and extent of absorption of SHR2554 following single oral doses of SHR2554 by assessment of maximum plasma concentration. | PK samples collected in both period 1 and 2 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post SHR2554 dose
AUC0-t of SHR2554: Assessment of the PK of SHR2554 using area under the plasma concentration curve from zero extrapolated to o the time of the last quantifiable concentration. | PK samples collected in both period 1 and 2 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post SHR2554 dose
AUC0-∞ of SHR2554: Assessment of the PK of SHR2554 using area under the plasma concentration-time curve from zero to infinity. | PK samples collected in both period 1 and 2 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post SHR2554 dose
Tmax of SHR2554: Assessment of the PK of SHR2554 using time to reach maximum plasma concentration. | PK samples collected in both period 1 and 2 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post SHR2554 dose
t1/2 of SHR2554: Assessment of the PK of SHR2554 using the terminal half-life. | PK samples collected in both period 1 and 2 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post SHR2554 dose
CL/F of SHR2554: Assessment of the PK of SHR2554 using the apparent plasma clearance. | PK samples collected in both period 1 and 2 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post SHR2554 dose
Vz/F of SHR2554: Assessment of the PK of AZD9291 using the apparent volume of distribution. | PK samples collected in both period 1 and 2 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, and 48 hours post SHR2554 dose

SECONDARY OUTCOMES:
Incidence and severity of adverse events/serious adverse events | From Day 1 to Day 15
Change in Fridericia-corrected QTc interval (QTcF) relative to baseline (ΔQTcF) | ECG samples collected in period 1 at pre-dose,1, 2, 3, 4, 6, 8, 12, and 24 hours post SHR2554 dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided